CLINICAL TRIAL: NCT01437631
Title: Does a Prophylactic Clip Application Decrease IPPB(Immediate Postpolypectomy Bleeding) and DPPB(Delayed Postpolypectomy Bleeding) After Colonoscopic Removal for a Large Pedunculated Polyps (>1cm)?
Brief Title: EFficacy of Prophylactic Clip Application in Decrease of Immediate Postpolypectomy Bleeding and Delayed Postpolypectomy Bleeding After Colonoscopic Removal for a Large Pedunculated Polyps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Kyung-Jo Kim, Clinical Associate Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2011-0653
Record Dates: First submitted 2011-09-19; First posted 2011-09-21 (Estimated); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Polyp of Large Intestine
Keywords: colon polyp; endoscopic polypectomy; postpolypectomy bleeding; prophylactic clip application
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- endoclip (Experimental): The group of patients who undergo prophylactic clip application after colonoscopic polypectomy of a large pedunculated polyp(>1cm).
  Interventions: Procedure: prophylactic clip application
- no endoclip (No Intervention): The group of patients who do not undergo prophylactic clip application after colonoscopic polypectomy of a large pedunculated polyp(>1cm).

INTERVENTIONS:
Procedure: prophylactic clip application — prophylactic clip application after colonoscopic polypectomy
  Arms: endoclip

SUMMARY:
The aim of this study is to evaluate the efficacy of prophylactic clip application after colonoscopic removal for a large pedunculated polyp (> 1cm) in preventing immediate postpolypectomy bleeding (IPPB) and delayed postpolypectomy bleeding (DPPB).

ELIGIBILITY:
Inclusion Criteria:

* Patients who have a large pedunculated polyp(>1cm) in the colon

Exclusion Criteria:

* Age under 20 years
* Subjects who are taking anticoagulants
* Subjects who have an abnormal coagulogram (platelet count, international normalized ratio, or activated partial thromboplastin time)
* Subjects who have inflammatory bowel diseases

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2011-09-01; Primary Completion 2015-04-30 (Actual); Study Completion 2015-04-30 (Actual)

PRIMARY OUTCOMES:
the occurrence of immediate post-polypectomy bleeding | 1 day
  At 1 day after endoscopic polypectomy, CBC will be done.
the occurrence of delayed post-polypectomy bleeding | 2 weeks
  At 2 weeks after endoscopic polypectomy, history of hematochezia will be taken at outpatient clinic.

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Jo Kim, M.D., Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Background] Shioji K, Suzuki Y, Kobayashi M, Nakamura A, Azumaya M, Takeuchi M, Baba Y, Honma T, Narisawa R. Prophylactic clip application does not decrease delayed bleeding after colonoscopic polypectomy. Gastrointest Endosc. 2003 May;57(6):691-4. doi: 10.1067/mge.2003.193. PMID 12709699
- [Derived] Soh JS, Seo M, Kim KJ. Prophylactic clip application for large pedunculated polyps before snare polypectomy may decrease immediate postpolypectomy bleeding. BMC Gastroenterol. 2020 Mar 12;20(1):68. doi: 10.1186/s12876-020-01210-5. PMID 32164613